CLINICAL TRIAL: NCT01499121
Title: A Phase II, Multi-Centre, Study of the Efficacy and Safety of Sunitinib Given on an Individualized Schedule as First-Line Therapy for Metastatic Renal Cell Cancer
Brief Title: Study of Efficacy and Safety of Sunitinib Given on an Individualized Schedule
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Dr. Georg Bjarnason, Medical Oncologist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OZM-042
Record Dates: First submitted 2011-12-12; First posted 2011-12-26 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Clear Cell, Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sunitinib (Other): Starting dose/schedule of Sunitinib 50 mg/28 days on, 14 days off. The intent is to maximize dose intensity of Sunitinib and minimize time off therapy based on individual tolerability using dose modification criteria.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — The starting dose will be 50 mg Sunitinib on the 28/14 schedule. In patients that develop ≥ grade-2 toxicity after 2 weeks, therapy will be held for 7 days or resolution before continuing therapy according to the 1st dose/schedule change. In patients that do not develop ≥ grade-2 toxicity, therapy will continue for 1-2 weeks or until ≥ grade-2 toxicity. In patients that develop > grade-2 toxicity after less than 4 weeks, therapy will be held for 7 days or before continued according to the 1st dose/schedule change. Patients that do develop grade-2 toxicity (but no more) on the 50 mg 28/14 schedule, will remain on schedule but the time off therapy will be reduced to 7 days if toxicity has resolved after a 7-day break. Patients that develop ≤ grade-1 toxicity on the 50 mg 28/14 schedule, will be dose escalated according to protocol.
  Other Names: Sutent; SU11248

SUMMARY:
This prospective single arm study will evaluate the efficacy and safety of sunitinib given on an individualized dosing schedule as first-line therapy in subjects with metastatic clear cell renal cell cancer. The treatment schedule intent is to maximize dose intensity of sunitinib and minimize time off therapy based on individual tolerability using protocol directed dose modification criteria. A total of 110 subjects will be enrolled. All subjects will continue to receive study treatment until disease progression or withdrawal of consent. The primary outcome for this study is progression-free survival (PFS), defined as the duration from the date a patient first receives Sunitinib until the date of death or confirmed progression according to the RECIST criteria.

DETAILED DESCRIPTION:
This is a single-arm, single-stage phase II study investigating the use of an individualized dosing regimen of Sunitinib on patients with metastatic renal cell carcinoma. The intent is to maximize dose intensity of sunitinib and minimize time off therapy based on individual tolerability using protocol directed dose modification criteria. Dose and schedule changes are done if toxicity (hematological, fatigue, skin, GI) is > grade 2. There will be no dosing or schedule changes for hypertension, hypothyroidism, skin color changes, heartburn, etc. unless clinically indicated. Subjects will continue therapy until progression according to RECIST 1.1 criteria. All subjects will be followed for progression free survival until progression but after 2 years on therapy, only grade 3/4 drug related adverse events will be recorded.

Fact-G and FKSI-DRS will be used to evaluate PRO/QOL at baseline and every 2 months timepoints. A more detailed pharmacokinetic blood sampling will be done in a subset of patients in an effort to understand if Sunitinib blood concentration has a tendency to go down during treatment, as has been shown to be the case for Sorafenib. Biomarker and genomics blood sampling for correlation with progression free survival, toxicity and pharmacokinetics will be collected at baseline and stored.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally recurrent or metastatic renal cell carcinoma of clear cell origin or with a component of clear cell histology.
* Patients with nephrectomy (partial or total) or without nephrectomy are eligible.
* Evidence of measurable disease by RECIST criteria version 1.1.
* Male or female, age ≥ 18 years old
* Karnofsky performance status ≥ 80 %.
* Adequate organ functions determined by protocol directed lab values
* Subject's willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Renal cell carcinoma without any clear (conventional) cell component.
* Prior systemic therapy of any kind for advanced RCC (including targeted therapy, immunotherapy, chemotherapy, hormonal, or investigational therapy). Prior neo-adjuvant or adjuvant therapy with cytokines, IL-2 or vaccines is only permitted if it did not occur within the preceding 12 months. Prior and/or concurrent bisphosphonate therapy is allowed.
* Major surgery or radiation therapy within 4 weeks of starting the study treatment. Prior palliative radiotherapy to metastatic lesion(s) is permitted, provided there is at least one measurable lesion that has not been irradiated
* NCI CTCAE Version 3.0 grade 3 haemorrhage within 4 weeks of starting the study treatment
* Diagnosis of any second malignancy within the last 5 years, except for adequately treated basal cell carcinoma, squamous cell skin cancer, or in situ cervical cancer
* Known brain metastases, spinal cord compression, or evidence of symptomatic brain or leptomeningeal carcinomatosis on screening CT or MRI scan.
* Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism
* Ongoing cardiac dysrhythmias of NCI CTCAE Version 3.0 grade ≥2
* Prolonged QTc interval on baseline EKG (>450 msec for males or >470 msec for females).
* Atrial Fibrillation of any grade.
* Uncontrolled hypertension (>150/100 mm Hg despite optimal medical therapy.
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness or other active infection.
* Concurrent treatment on another clinical trial. Supportive care trials or non-treatment trials, e.g. QOL, and imaging trials are allowed.
* Concomitant treatment with a drug having proarrhythmic potential
* Use of potent CYP3A4 inhibitors and inducers 7 and 12 days before dosing, respectively
* Pregnancy or breastfeeding. Female subjects must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of therapy. All female subjects with reproductive potential must have a negative pregnancy test (serum) prior to enrolment. Male subjects must be surgically sterile or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2012-05; Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Progression free survival for sunitinib given on an individualized dose/schedule | 3.5 years
  Primary objective is to characterize the progression free survival for sunitinib given on an individualized dose/schedule in patients on first-line treatment for metastatic renal cell cancer. Subjects will continue therapy until progression according to RECIST criteria version 1.1. Tumour measurements using physical exam, spiral CT scan and/or MRI or other appropriate techniques deemed suitable by the investigator will be performed at screening and repeated at the end of every 2 cycles until disease progression.

SECONDARY OUTCOMES:
Patient tolerability and safety of an individualized dose/schedule | 3.5 years
  To evaluate the tolerability and safety of individualized dose/schedule changes and dose escalation and schedule modification in patients with minimal toxicity after treatment with sunitinib 50 mg for 28 days. The adverse effects of the drug will be assessed from adverse events, vital signs and by clinically significant changes in the lab evaluations and ECG's. Categorical endpoints, will be summarized using proportions and frequencies.
Dose intensity of sunitinib given on an individualized dose/schedule. | 3.5 years
  The intent is to maximize dose intensity of sunitinib and minimize time off therapy based on individual tolerability using the dose modification criteria outlined in the protocol. Dose and schedule changes are done if toxicity (hematological, fatigue, skin, GI) is > NCI CTCAE (version 3) grade 2. Patients that tolerate the standard 50 mg 28 days on/14 days off schedule with minimal toxicity (grade 1) will be dose escalated in 12.5 mg increments as outlined in the protocol on a schedule of 14 days on and 7 days off to a maximum of 75 mg.
Overall survival and patient quality of life | 3.5 years
  To characterize the overall survival and study the quality of life in subjects given sunitinib on an individualized dose/schedule. Quality of life questionnaires (ie. FACT-G and FKSI-DRS) will be completed at baseline and every 2 months thereafter until disease progression. Summary scores for QOL outcomes will be reported as the raw value at each time point evaluated, as well as the change in score from baseline. Overall survival will be calculated from the date of registration and estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Georg A. Bjarnason, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (13):
- Canada (13):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Agency - Vancouver, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Kingston General Hospital Research Institute, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Durham Regional Cancer Centre, Oshawa, Ontario
  - Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Notre-Dame Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Bjarnason GA, Knox JJ, Kollmannsberger CK, Soulieres D, Ernst DS, Zalewski P, Canil CM, Winquist E, Hotte SJ, North SA, Heng DYC, Macfarlane RJ, Venner PM, Kapoor A, Hansen AR, Eigl BJ, Czaykowski P, Boyd B, Wang L, Basappa NS. The efficacy and safety of sunitinib given on an individualised schedule as first-line therapy for metastatic renal cell carcinoma: A phase 2 clinical trial. Eur J Cancer. 2019 Feb;108:69-77. doi: 10.1016/j.ejca.2018.12.006. Epub 2019 Jan 14. PMID 30648632